CLINICAL TRIAL: NCT03111511
Title: A Phase 1, Open-label Study in Healthy Female Subjects to Investigate the Effect of JNJ-56136379 at Steady-state on the Single-dose Pharmacokinetics of Ethinylestradiol and Drospirenone (Oral Contraceptive) and on the Single-dose Pharmacokinetics of Midazolam (Probe Substrate for Cytochrome P450 3A4)
Brief Title: A Study in Healthy Female Participants to Investigate the Effect of JNJ-56136379 at Steady-state on the Single-dose Pharmacokinetics of Ethinylestradiol and Drospirenone (Oral Contraceptive) and on the Single-dose Pharmacokinetics of Midazolam (Probe Substrate for Cytochrome P450 3A4)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR108309; 56136379HPB1004 (Other: Janssen Sciences Ireland UC); 2017-000365-70 (EudraCT Number)
Record Dates: First submitted 2017-03-20; First posted 2017-04-12 (Actual); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Healthy
MeSH Terms: interventions — drospirenone; Ethinyl Estradiol; drospirenone and ethinyl estradiol combination; Midazolam; JNJ-56136379

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Drospirenone/Ethinylestradiol + Midazolam + JNJ-56136379 (Experimental): Participants will receive single dose of drospirenone/ethinylestradiol 3 milligram (mg)/0.02 mg (oral contraceptive [OC]) and single dose of midazolam 2 mg under fasted conditions on Day 1. JNJ-56136379 250 mg twice daily will be administered on Days 6, 7 and JNJ-56136379 170 mg once daily on Days 8 to 25 under fed conditions, except on Day 21 on which Single dose of JNJ-56136379 170 mg + single dose of OC and single dose of midazolam 2 mg will be administered on fasted state. A single dose of drospirenone/ethinylestradiol 3 mg/0.02 mg and midazolam 2 mg on Day 21 under fasted conditions.
  Interventions: Drug: Drospirenone/Ethinylestradiol; Drug: Midazolam; Drug: JNJ-56136379

INTERVENTIONS:
Drug: Drospirenone/Ethinylestradiol — A single dose of drospirenone/ethinylestradiol 3 mg/0.02 mg (OC) tablets on Days 1 and 21.
  Other Names: Betadex clathrate (Yaz)
Drug: Midazolam — Midazolam 2 mg orally on Days 1 and 21.
Drug: JNJ-56136379 — JNJ-56136379 dose will be administered orally at a dose of 250 mg (as 2 tablets of 100 mg + 2 tablets of 25 mg) on Days 6 and 7 and at a dose of 170 mg (as 1 tablet of 100 mg+ 2 tablets of 25 mg + 4 tablets of 5 mg) on Days 8 to 25.

SUMMARY:
The main purpose of this study is to evaluate the effect of steady-state concentrations of JNJ-56136379 on the single-dose pharmacokinetics (PK) of drospirenone and ethinylestradiol (oral contraceptive [OC]) in healthy female participants and to evaluate the effect of steady-state concentrations of JNJ-56136379 on the single-dose PK of midazolam (sensitive probe substrate for CYP3A4) in healthy female participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, and vital signs performed at screening. If there are abnormalities, the participant may be included only if the investigator judges the abnormalities to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* healthy on the basis of clinical laboratory tests performed at screening
* must have a normal 12-lead electrocardiogram (ECG) at screening including: normal sinus rhythm (heart rate between 45 and 100 beats per minute [bpm], extremes included); QT interval corrected for heart rate (QTc) according to Fridericia (QTcF) less than equal to (<=)470 milliseconds (ms); QRS interval less than (<)120 ms; PR interval <=220 ms
* must have a blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeters of mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic. If blood pressure is out of range, up to 2 repeated assessments are permitted
* must have a body mass index (BMI; weight in kg divided by the square of height in meters) between 18.0 and 30.0 kilogram per square meter (kg/m^2), extremes included, and a body weight not less than 50.0 kilogram (kg)

Exclusion Criteria:

* any evidence of heart block or bundle branch block
* history of liver or renal dysfunction (estimated creatinine clearance <60 milliliters per minute (mL/min) at screening, calculated by the Modification of Diet in Renal Disease [MDRD] formula12), significant cardiac, vascular, pulmonary, gastrointestinal (such as significant diarrhea, gastric stasis, or constipation that in the investigator's opinion could influence drug absorption or bioavailability), endocrine, neurologic, hematologic, rheumatologic, psychiatric, neoplastic, or metabolic disturbances
* past history of cardiac arrhythmias (example [eg], extrasystoli, tachycardia at rest), history of risk factors for Torsade de Pointes syndrome (eg, hypokalemia, family history of long QT Syndrome)
* current human immunodeficiency virus type 1 (HIV-1) or HIV-2 infection (confirmed by antibodies) at screening
* any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, and urticaria

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-08-23 (Actual); Study Completion 2017-08-23 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration of Drospirenone (Cmax) | Day 1 and 21: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12 hours postdose
  The Cmax is the maximum observed plasma analyte concentration.
Area Under the Analyte Concentration-time Curve From Time Zero to the Time of the Last Measurable Concentration of Drospirenone (AUC [0-last]) | Day 1 and 21: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12 hours postdose
  The AUC (0-last) is the area under the analyte concentration-time curve from time 0 to time of the last quantifiable concentration.
Area Under the Analyte Concentration-time Curve From Time Zero to Infinite Time of Drospirenone (AUC [0-infinity]) | Day 1 and 21: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12 hours postdose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Maximum Observed Plasma Concentration of Ethinylestradiol (Cmax) | Day 1 and 21: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12 hours postdose
  The Cmax is the maximum observed plasma analyte concentration.
Area Under the Analyte Concentration-time Curve From Time Zero to the Time of the Last Measurable Concentration of Ethinylestradiol (AUC [0-last]) | Day 1 and 21: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12 hours postdose
  The AUC (0-last) is the area under the analyte concentration-time curve from time 0 to time of the last quantifiable concentration.
Area Under the Analyte Concentration-time Curve From Time Zero to Infinite Time of Ethinylestradiol (AUC [0-infinity]) | Day 1 and 21: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12 hours postdose
  The AUC (0-infinity) is the area under the analyte concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the analyte concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Maximum Observed Plasma Concentration of Midazolam and its Metabolite 1-OH-Midazolam (Cmax) | Day 1 and 21: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 9, 12 hours postdose on Day 1
  The Cmax is the maximum observed plasma analyte concentration.
Area Under the Analyte Concentration-time Curve From Time Zero to Infinite Time of Midazolam and its Metabolite 1-OH-Midazolam (AUC [0-infinity]) | Day 1 and 21: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 9, 12 hours postdose
  The AUC (0-infinity) is the area under the analyte concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the analyte concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.
Area Under the Analyte Concentration-time Curve From Time Zero to the Time of the Last Measurable Concentration of Midazolam and its Metabolite 1-OH-Midazolam (AUC [0-last]) | Day 1 and 21: 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 9, 12 hours postdose
  The AUC (0-last) is the area under the analyte concentration-time curve from time 0 to time of the last quantifiable concentration.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Up to 30-35 days after last study drug administration (approximately 70 days)
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Maximum Observed Plasma Concentration of JNJ-56136379 (Cmax) | 1, 2, 4, 9 and 12 hours postdose on Day 21
  The Cmax is the maximum observed plasma analyte concentration.
Area Under the Concentration-time Curve From Time Zero to tau Hours Postdose of JNJ-56136379 (AUCtau) | Predose, 1, 2, 4, 9 and 12 hours postdose on Day 21; predose on Day 22
  AUCtau is area under concentration-time curve from time 0 to tau hours postdose, calculated by linear-linear trapezoidal summation.
Steady-state Plasma Concentration of JNJ-56136379 After Multiple Dosing | Days 16, 19, 20 and 21 (predose)
  Steady-state plasma concentration of JNJ-56136379 will be evaluated after multiple dosing.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium